CLINICAL TRIAL: NCT05715892
Title: An Observational Study Investigating The Experiences of Patients In Gastric Bypass Clinical Trials
Brief Title: Examining Patterns in the Involvement of Gastric Bypass Patients in Clinical Studies
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80772648
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Gastric Bypass; Weight Loss Surgery
Keywords: gastric bypass; weight loss surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trial participation has historically been heavily biased toward specific demographics.

Several people will be invited to enroll in this study so that it may collect a variety of data about gastric bypass clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

The information collected from this study can be used to improve patient experience and outcomes for future patients and an opportunity to contribute to the advancement of medical knowledge and treatments for gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of obesity or disorder of metabolism undergoing routine gastric bypass surgical intervention
* Capable of giving signed informed consent.

Exclusion Criteria:

* ECOG score of 4
* Ineligible for gastric bypass surgery
* Pregnant women or women actively seeking to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric bypass patients who are actively considering participating in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a gastric bypass clinical study | 3 months
Rate of gastric bypass patients who remain until trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982
- [Background] Fisher BL, Barber AE. Gastric bypass procedures. Eur J Gastroenterol Hepatol. 1999 Feb;11(2):93-7. doi: 10.1097/00042737-199902000-00007. PMID 10102217
- [Background] Collins BJ, Miyashita T, Schweitzer M, Magnuson T, Harmon JW. Gastric bypass: why Roux-en-Y? A review of experimental data. Arch Surg. 2007 Oct;142(10):1000-3; discussion 1004. doi: 10.1001/archsurg.142.10.1000. PMID 17938315

DOCUMENTS (1):
  • Informed Consent Form (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT05715892/ICF_000.pdf